CLINICAL TRIAL: NCT05703919
Title: Standard vs Targeted Oxygen Therapy Prehospital for Chronic Obstructive Pulmonary Disease
Acronym: STOP-COPD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5925; 2022-502003-30-00 (Other: https://euclinicaltrials.eu)
Record Dates: First submitted 2023-01-10; First posted 2023-01-30 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: COPD Exacerbation; COPD Exacerbation Acute
Keywords: Titrated Oxygen; COPD Exacerbation; Prehospital; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, randomized 1:1, parallel groups, patient blinded, prehospital, single center, acute, superiority trial
Who Masked: Participant
Masking Description: The trial will be single blinded. The patients will be blinded to treatment allocation. The EMTs (emergency medical technicians) or paramedics will not be blinded because of practical, ethical and security problems with carrying compressed gas without known content in an ambulance. As part of study informed and training, the EMT's and paramedics will be attentive to keep all AECOPD suspected patients blinded to the treatment allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titrated Oxygen (Experimental): If the treating EMT or paramedic finds indications for inhaled bronchodilators, this will be done with compressed air 6-8 l/min. as the driver for the nebulizer. The patient will have a Bi-nasal EtCO2 (end-tidal carbon dioxide) meter placed under the nebulizer. This will measure the EtCO2 during the treatment and at the same time oxygen can be titrated through this to a target SpO2 of 88-92%. Repeated treatment will be at the discretion of the treating EMT or paramedic according to SOP (standard operating procedures).
  Following scenarios regarding SpO2 can occur during treatment:
  SpO2 <88%: Supplemental oxygen via the EtCO2-meter up to 10 l/min, if higher oxygen levels are needed oxygen will be used as driver for the nebulizer. If the SpO2 remains under 88% additional oxygen can be added via the EtCO2-meter.
  SpO2 88-92%: No intervention.
  SpO2 >92%: No intervention.
  If repeated treatment is not indicated the patient receives oxygen to SpO2 88-92% according SOP.
  Interventions: Drug: Titrated Oxygen
- Standard Oxygen (Active Comparator): If the treating EMT or paramedic finds indication for inhaled bronchodilators, this will be done with oxygen 6-8 l/min. as the driver for the nebulizer. The patient will have a Bi-nasal EtCO2 meter placed under the nebulizer. This will measure the EtCO2 during the treatment and at the same time mask the patient for group allocation. Repeated treatment will be at the discretion of the treating EMT or paramedic according to SOP.
  Following scenarios regarding SpO2 can occur during treatment:
  SpO2 <88%: Supplemental oxygen via the EtCO2 -meter up to 10 l/min.
  SpO2 88-92%: No intervention.
  SpO2 >92%: No intervention.
  If repeated treatment is not indicated the patient receives oxygen to SpO2 88-92% according SOP.
  Interventions: Drug: Standard Oxygen

INTERVENTIONS:
Drug: Titrated Oxygen — Titrated oxygen strategy - a mix of supplemental oxygen and compressed atmospheric air as driver for inhaled bronchodilators to target SpO2 88-92%
  Other Names: Oxygen titration to SpO₂ 88-92% and compressed atmospheric air as nebulizer driver
  Arms: Titrated Oxygen
Drug: Standard Oxygen — Standard care using compressed oxygen (100%) as driver for inhaled bronchodilators
  Other Names: No SpO₂ target restriction and 100% compressed oxygen as nebulizer driver
  Arms: Standard Oxygen

SUMMARY:
The STOP-COPD trial is a randomized, patient-blinded, prehospital clinical trial designed to evaluate the effect of titrated oxygen therapy compared to standard oxygen treatment in patients with suspected acute exacerbation of chronic obstructive pulmonary disease (AECOPD) treated with inhaled bronchodilators. The primary objective is to determine whether a titrated oxygen strategy targeting SpO₂ 88-92% can reduce 30-day mortality compared to the current standard practice using 100% compressed oxygen as a nebulizer driver.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a leading cause of morbidity and mortality globally. In the prehospital setting, patients with suspected acute exacerbation of COPD (AECOPD) are frequently treated with inhaled bronchodilators driven by 100% oxygen, despite concerns that high-concentration oxygen therapy may worsen hypercapnia and acidosis, leading to increased mortality.

The STOP-COPD trial is a prospective, randomized, parallel-group, superiority trial conducted in the Prehospital Emergency Medical Services, Central Denmark Region. Patients aged 40 years or older with suspected AECOPD requiring inhaled bronchodilators are randomized 1:1 to receive either:

Titrated oxygen therapy: Inhaled bronchodilators driven by compressed air with supplemental oxygen titrated to maintain SpO₂ 88-92%.

Standard treatment: Inhaled bronchodilators driven by 100% compressed oxygen according to standard protocols.

The primary outcome is 30-day all-cause mortality. Secondary outcomes include 24-hour and 7-day mortality, need for invasive or non-invasive ventilation, development of respiratory acidosis upon hospital arrival, ICU admission rate, length of hospital and ICU stay, patient-experienced dyspnoea, and readmission rates. A total of 1,888 patients will be enrolled.

The study is conducted under emergency research regulations allowing enrolment before informed consent, with consent obtained as soon as feasible after hospital admission. This trial seeks to evaluate whether titrating oxygen delivery in the prehospital phase can improve survival and clinical outcomes for patients with AECOPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 40
* EMT or Paramedic suspected AECOPD
* Confirmed suspicion of COPD

Exclusion Criteria:

* Bronchospasm due to asthma, allergic reaction or non-COPD conditions
* Known or suspected pregnancy
* Prehospital Non-invasive, invasive or assisted bag mask ventilation
* Allergy to inhaled bronchodilators (Salbutamol)
* Inter-hospital transfer
* More than 2 doses (5 mg salbutamol) inhalation drug, acute treatment by EMS (emergency medical service) personnel, before allocated treatment is initiated
* Suspicion of acute coronary syndrome

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1888 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Mortality, 30-day | Day 30 from randomization
  Vital status assessed 30 days after randomization using hospital electronic medical records

SECONDARY OUTCOMES:
Mortality, 24-hour | 24 hours from randomization
  Vital status assessed 24 hours after randomization using hospital electronic medical records
Mortality, 7-day | Day 7 from randomization
  Vital status assessed 7 days after randomization using hospital electronic medical records
Length of hospital stay | Day 30 from randomization
  Number of days from hospital admission to hospital discharge, collected from hospital electronic medical records
ICU admission rate | Day 30 from randomization
  Proportion of patients admitted to an intensive care unit during the index hospitalization, collected from the electronic hospital medical record
Length of ICU stay | Day 30 from randomization
  Number of days spent in the intensive care unit during the index hospitalization, collected from the patient's electronic hospital medical record
In-hospital need for NIV (non-invasive ventilation) within 24 hours | Day 30 from randomization
  Use of non-invasive ventilation recorded within 24 hours of hospital admission, collected from the patient's electronic hospital medical record
In-hospital need for NIV within 7 days | Day 30 from randomization
  Use of non-invasive ventilation recorded within 7 days of hospital admission, collected from the patient's electronic hospital medical record
In-hospital need for NIV within 30 days | Day 30 from randomization
  Use of non-invasive ventilation recorded within 30 days of randomization, collected from the patient's electronic hospital medical record
Time to NIV | Day 30 from randomization
  Time from hospital admission to initiation of non-invasive ventilation, collected from the patient's electronic hospital medical record
In-hospital need for invasive mechanical ventilation within 24 hours | Day 30 from randomization
  Initiation of invasive mechanical ventilation within 24 hours of hospital admission, collected from the patient's electronic hospital medical record
In-hospital need for invasive mechanical ventilation within 7 days | Day 30 from randomization
  Initiation of invasive mechanical ventilation within 7 days of hospital admission, collected from the patient's electronic hospital medical record
In-hospital need for invasive mechanical ventilation within 30 days | Day 30 from randomization
  Initiation of invasive mechanical ventilation within 30 days of randomization, collected from the patient's electronic hospital medical record
Time to invasive ventilation | Day 30 from randomization
  Time from hospital admission to initiation of invasive mechanical ventilation, collected from the patient's electronic hospital medical record
Proportion of patients with respiratory acidosis on arrival to hospital | Day 30 from randomization
  Presence of respiratory acidosis (PaCO₂ >6.3 kPa and pH <7.35) assessed via arterial blood gas analysis within 30 minutes after arrival, collected from the patient's electronic hospital medical record
The degree of acidosis based on the pH (potential of hydrogen) value | Day 30 from randomization
  Lowest pH value measured from arterial blood gas within 30 minutes of hospital arrival, collected from the patient's electronic hospital medical record
Patient experienced dyspnoea on a verbal rating scale 0-10 | Day 30 from randomization
  Patient-reported dyspnoea score at hospital arrival on a scale from 0 (no dyspnoea) to 10 (worst imaginable dyspnoea), collected from the prehospital patient record and hospital medical record
Readmission rate | Day 30 after discharge
  Proportion of patients readmitted to hospital within 30 days after discharge from index hospitalization, collected from the patient's electronic hospital medical record
Time to readmission | Day 30 after discharge
  Number of days from hospital discharge to first hospital readmission within 30 days, collected from the patient's electronic hospital medical record

CONTACTS AND LOCATIONS:
Overall Officials: Martin F Gude, PhD, Principal Investigator — Central Denmark Region
Locations (1):
- Prehospital Emergency Medical Servises, Central Denmark Region, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available to researchers whose proposed use of the data has been approved by the local administration. Data will be shared starting 9 months after publication of the primary results and will be accessible until data are no longer stored, according to current ICMJE recommendations and EU data protection regulations.
  All trial-related documents (e.g., protocol, statistical analysis plan) will be made publicly available on the trial website. Patient-related data will not be accessible on the website.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 9 months after primary results publication; data will remain available until de-identified data are no longer stored according to ICMJE recommendations and EU regulations.
Access Criteria: Researchers must submit a methodologically sound proposal for use of the data. Access will be granted following review and approval by the local trial administration. A data-sharing agreement will be required.
URL: http://www.STOP-COPD.com

REFERENCES:
- [Derived] Jensen ASR, Valentin JB, Mulvad MG, Hagenau V, Skaarup SH, Johnsen SP, Vaeggemose U, Gude MF. Standard vs. targeted oxygen therapy prehospitally for chronic obstructive pulmonary disease (STOP-COPD): study protocol for a randomised controlled trial. Trials. 2024 Jan 25;25(1):85. doi: 10.1186/s13063-024-07920-5. PMID 38273393

DOCUMENTS (2):
  • Study Protocol (2025-05-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT05703919/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT05703919/SAP_001.pdf